CLINICAL TRIAL: NCT07270510
Title: Clinical and Volumetric Evaluation of Collagen Matrix Efficacy in Alveolar Socket Preservation, Randomized Clincal Trial
Brief Title: The Effect of Collagen In Tooth Extraction Procedures
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Altinbas University (Other)
Responsible Party: Principal Investigator, Gulhuseyn Abdullayev, Dr., Altinbas University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025/136 REV2
Record Dates: First submitted 2025-11-26; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Extraction Socket Healing; Extraction, Tooth
Keywords: collagen matrix; alveolar socket preservation; alveolar ridge; bone resorption; socket seal
MeSH Terms: conditions — Bone Resorption

STUDY DESIGN:
Intervention Model Description: The study is a parallel arm randomized clinical trial consisting of a control and a test group with same number of participants.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor was blinded to minimize data analysis bias..
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (No Intervention): The control group only went through routine tooth extractions without further interventions. Extraction sockets were left to spontaneous healing.
- Test Group (Active Comparator): The test group received Collagen Matrix onto their extraction sockets after extractions.
  Interventions: Device: Collagen Matrix soft tissue graft

INTERVENTIONS:
Device: Collagen Matrix soft tissue graft — Circular 8 mm diameter collagen matrix grafts were sutured to seal extraction sockets in the participants. The sutures were removed 1 week after the intervention.
  Arms: Test Group

SUMMARY:
This study is aimed at assessing the effect of an animal-derived collagen matrix on bone and soft tissues in the human teeth. Single-rooted teeth that are beyond restoration and in need of extraction will be included in the study. Patients will be divided into two comparable groups in a randomized manner. The first group will proceed with tooth extraction only, which will be left for spontaneous healing. The second (test) group will receive an additional collagen matrix graft after the extraction, which will be sutured to the tooth socket. Sutures will be removed 1 week after surgery. Both groups will undergo CBCT imaging on the day of surgery and at the 3-month follow-up. Differences in bone measurements like height and width will be recorded as well as soft tissue measurements like thickness and width. Data acquired from two groups will be compared against each other to specify the protective effect of the applied collagen matrix graft.

DETAILED DESCRIPTION:
To assess the clinical and volumetric efficacy of the porcine-derived collagen matrix during alveolar socket preservation is aimed in this study that is a randomized controlled clinical trial including two study groups. 24 participants with extraction indication in their non-molar teeth that are eligible will be recruited to the study according to the inclusion criteria of the trial. After the initial oral assessment, the participants were allocated into one of the groups via online randomizer software. Both groups will have the teeth extracted in an atraumatic way using dental periotomes to reduce the surgical trauma and unfavorable healing pattern. Control group sockets will heal spontaneously without any additional procedures. Test group sockets will be applied 8 mm circular collagen matrix grafts with 5/0 propylene sutures to secure the grafts in the sockets. The sutures will be removed at the 1-week follow-up. Both groups will be prescribed analgesic drugs and antimicrobial oral rinse. CBCT imaging will be performed right after surgery and at the 3-month follow-up. Volumetric measurements, like bone heights and widths, will be recorded in this period. Soft tissue changes will be recorded by oral examinations. Inter-group and intra-group differences will be assessed statistically.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults (absence of cardiovascular diseases, thyroid diseases, oncological diseases Non-smokers Extraction diagnosis on non-molar teeth Gingivitis, stage 1-2 periodontitis conditions Absence of radiotherapy last 2 years Non restorable teeth (deep fracture, excessive caries, failed root canal treatment) Overall plaque score and gingival score of <10%

Exclusion Criteria:

Systemically compromised patients Smokers Pregnancy or lactation Heavy periodontally compromised patients (Stage 3-4) Patients undergone radiotherapy in the last 2 years Collagen allergic patients Restorable teeth Overall plaque score and gingival score of >10%

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
Buccal Height (BH) | From intervention day to 3 months follow-up
  Measurement of Buccal Height using CBCT scans
Buccal Width (BW) | From intervention day to 3-month follow-up
  Buccal Width measurements using CBCT scans

SECONDARY OUTCOMES:
Palatal/lingual Height (PH) | From intervention day to 3-month follow-up
  Palatal/lingual height measuerements using CBCT scans
Palatal/lingual Width (PW) | From intervention day to 3-month follow-up
  Palatal/lingual width measurements using CBCT scans
Gingival Thickness (GT) | From intervention day to 3-month follow-up
  Gingival Thickness measurement using periodontal probe
Keratinized Tissue Width (KTW) | From intervention day to 3-month follow-up
  Keratinized Tissue Width measured using periodontal probe

CONTACTS AND LOCATIONS:
Overall Officials: Sebnem Dirikan Ipci, Prof., Study Director — Altinbas University
Locations (1):
- Altinbas University, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
IPD sharing may be available upon rasonable request

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-11-26): https://cdn.clinicaltrials.gov/large-docs/10/NCT07270510/Prot_SAP_000.pdf